CLINICAL TRIAL: NCT00733070
Title: A Multicenter Multinational Study to Evaluate the Safety and Efficacy of the CiTop™ ExPander™ Guidewire for Crossing Chronic Total Occlusions in Coronary Arteries
Brief Title: Study to Evaluate the Safety and Efficacy of the CiTop™ ExPander™ Guidewire for Crossing Chronic Total Occlusions in Coronary Arteries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no interest to develop the product
Sponsor: Ovalum (Industry)
Responsible Party: Nathalie Gilat, Ovalum
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OVC-003-00
Record Dates: First submitted 2008-08-10; First posted 2008-08-12 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Chronic Total Occlusion
Keywords: CTO; Chronic Total Occlusion; Revascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CiTop™ ExPander™ Guidewire — Chronic Total Occlusion guidewire

SUMMARY:
A multicenter multinational study to evaluate the safety and efficacy of the CiTop™ ExPander™ Guidewire for crossing chronic total occlusion in Coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained prior to any trial activities.
2. Patients, male or female between 21 and 80 years of age, with no significant co-morbidities (see exclusion criteria).
3. Patient has an angiographic documented Chronic Total Occlusion showing distal TIMI flow 0 to 1.

Exclusion Criteria:

1. Patient unable to give informed consent.
2. Current participation in another study with any investigational drug or device.
3. Factors making follow-up and/or repeat angiography difficult or unlikely.
4. Contra-indication to emergency artery by pass surgery.
5. Lack of surgical backup.
6. Contra-indication to treatment with Aspirin, or Clopidogrel and/or Heparin.
7. Lesion > 40mm in length (both calcified lesion and adjacent thrombus).
8. Treated vessel referenced diameter less than 2.5 mm.
9. Visualization of the distal lumen less than the Rentrop Classification Grade 2 collateralization.
10. Non-visible entry point of target lesion.
11. Totally occluded bypass graft as target vessel.
12. Acute MI less than 1 week before procedure.
13. Patient has significant LV dysfunction, 35% LVEF or less.
14. Patient with cancer or other sever chronic disease with life expectance of 2 years.
15. Patient has chronic renal failure with serum creatinine ≥2.
16. Hemoglobin ≤11.
17. Patient is known or suspected not to tolerate the contrast agent.
18. Morbid Obesity (BMI > 40).
19. Drug abuse or alcoholism.
20. Patients under custodial care.
21. Pregnant women or women with childbearing potential with a positive pregnancy test at the time of procedure.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Angiographic documentation of placement of CiTop™ distal to occlusion with no device related major complications | during procedure, 1day, 1week and 30 days post procedure

SECONDARY OUTCOMES:
Successful stenting | During procedure, Day1, Day7 and Day30 post procedure
Wire crossing duration | during procedure
Fluoroscopy time | during procedure
Amount of contrast | during procedure
Maneuverability of the CiTop™ up to the occlusion | during procedure
No mechanical damage to the device during | during procedure

CONTACTS AND LOCATIONS:
Locations (3):
- HELIOS Klinikum Wuppertal, Wuppertal, Germany
- South Africa (2):
  - Sunward Park Hospital, Boksburg
  - Sunninghill Hospital, Sunninghill